CLINICAL TRIAL: NCT07173114
Title: New Approaches for Evaluating the Interchangeability of Reference Materials and Quality Controls (COMET-MPL)
Acronym: COMET-MPL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0369
Record Dates: First submitted 2025-09-01; First posted 2025-09-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hospitalization; All Conditions
Keywords: In Vitro Diagnostics (IVD); Commutability; Calibration; Interchangeability; Analytical Validity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Recruiting a panel of fresh clinical samples with values close to those of standards or quality controls requires the collection of three 7 mL tubes of blood during a scheduled check-up as part of routine care. After centrifugation, the serum will be aliquoted and the samples sent to the various medical laboratories performing the assays for which commutability will be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Panel 1: Patients aged 18 years or older
- Panel 2: Patients aged 18 years or older receiving immunosuppressive therapy (cyclosporine and/or everolimus and/or tacrolimus and/or sirolimus)

SUMMARY:
Medical biology tests are essential to clinical decision-making. The European Regulation on in vitro diagnostic medical devices (EU/2017/746) requires metrological traceability of the values assigned to calibrators and quality controls, based on reference measurement methods (RMMs) or certified reference materials (CRMs). However, these references are not available for all analyses, limiting manufacturers' ability to comply with regulatory requirements.

The dissemination of traceability relies mainly on CRMs. However, to guarantee the validity of the results, these materials must have sufficient commutability, i.e., behavior comparable to that of native biological samples. This property is also required for external quality controls (EQA) used in external quality control programs. Commutability is an essential condition for avoiding matrix effects and ensuring the reliability of results.

The COMET-MPL project aims to optimize manufacturing processes for commutable, single-parameter, or multi-parameter CRMs and EQA. Evaluate the commutability of these materials in relation to patient samples.

The COMET-MPL project aims to Produce materials suitable for priority analyses: bilirubin, cyclosporine, parathyroid hormone (PTH), human cytomegalovirus, estradiol.

Commutability will be verified by comparing the performance of CRMs and EQA with that of clinical samples in several French laboratories equipped with automated systems from different manufacturers.

DETAILED DESCRIPTION:
The global in vitro diagnostics (IVD) market was valued at €91.1 billion in 2023 and is projected to reach €147.3 billion by 2030, reflecting its growing strategic importance in healthcare. Medical biology tests are central to clinical decision-making and must deliver reliable, accurate, reproducible, and standardized results across all medical laboratories.

Under Regulation (EU) 2017/746, the metrological traceability of values assigned to calibrators and quality control materials must be ensured through Reference Measurement Procedures (RMPs) and/or Certified Reference Materials (CRMs) of higher order. However, among the thousands of parameters routinely measured, fewer than 200 currently meet these requirements, making regulatory compliance difficult for IVD manufacturers and limiting laboratories' ability to meet ISO NF 15189 standards.

It is therefore essential to develop CRMs and External Quality Controls (EQA) that are compatible with high-throughput multiparameter analyzers used in medical laboratories. These materials must not only be traceable but also commutable, meaning they must behave similarly to native patient samples to ensure analytical validity.

The COMET-MPL project addresses this need by evaluating the interchangeability (commutability) of selected CRMs and EQA integrated into multiparametric preparations. These will be tested on automated high-throughput systems used in routine medical biology laboratories to assess their suitability as calibrators or quality controls under real-world conditions.

Each patient will participate in a single visit, during a scheduled blood draw as part of routine care. Three blood tubes will be collected, the serum will be aliquoted, and samples will be sent to partner laboratories for analysis.

The collective benefits of this study include:

* Improved patient care pathways, from initial diagnosis to therapeutic follow-up, through enhanced analytical quality of laboratory tests.
* Strengthened regulatory compliance for laboratories and IVD manufacturers.
* Availability of high metrological quality CRMs and EQA, facilitating alignment with ISO standards 15189.
* Greater reliability and comparability of biological results, contributing to more precise and equitable healthcare delivery.

ELIGIBILITY:
Inclusion Criteria:

* Panel 1: adults ≥ 18 years of age.
* Panel 2: adults ≥ 18 years of age undergoing immunosuppressive treatment (cyclosporine, everolimus, tacrolimus, sirolimus).

Exclusion Criteria:

* Protected patients (minors who are not emancipated, individuals who are unable to express their consent, etc.)
* Individuals who are not affiliated with a social security system
* Individuals under judicial protection
* Refusal to give consent to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of patients hospitalized in the departments of the investigative teams at Montpellier University Hospital, regardless of their pathologies.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Assessment of Commutability | 1 day
  The primary endpoint is the analytical data associated with the biomarker in question obtained from the blood sample: commutability will be assessed by comparing the behavior of certified reference materials (CRMs) and external quality controls (EQA) with the results from fresh serum.

SECONDARY OUTCOMES:
Serum Testosterone Concentration | 1 day
  Measured concentration (ng/dL) in patient serum samples using standardized laboratory methods
Serum Calcium Concentration | 1 day
  Measured concentration (mg/dL) in patient serum samples using standardized laboratory methods
Serum Glucose Concentration | 1 day
  Measured concentration (mg/dL) in patient serum samples using standardized laboratory methods
Total Cholesterol Concentration | 1 day
  Measured concentration (mg/dL) in patient serum samples using standardized laboratory methods
High-Density Lipoprotein Cholesterol (HDL-C) Concentration | 1 day
  Measured concentration (mg/dL) in patient serum samples using standardized laboratory methods
Triglyceride (TG) Concentration | 1 day
  Measured concentration (mg/dL) in patient serum samples using standardized laboratory methods
Alanine Aminotransferase (ALT) Activity | 1 day
  Measured concentration (U/L) in patient serum samples using standardized laboratory methods
Creatine Kinase (CK) Activity | 1 day
  Measured concentration (U/L) in patient serum samples using standardized laboratory methods
Serum Albumin Concentration | 1 day
  Measured concentration (g/dL) in patient serum samples using standardized laboratory methods
Non-commutability bias of certified reference materials (CRMs) consisting of Lyophilized serum spiked with exogenous compounds | 1 day
  measured (in %) by establishing difference plots between biochemical measurement results obtained for the CRMs and a panel of clinical specimens (see Clin Chem. 2018;64(3):455-464)
Non-commutability bias of certified reference materials (CRMs) consisting of Lyophilized serum not spiked with exogenous compounds | 1 day
  measured (in %) by establishing difference plots between biochemical measurement results obtained for the CRMs and a panel of clinical specimens (see Clin Chem. 2018;64(3):455-464)
Non-commutability bias of certified reference materials (CRMs) consisting of frozen serum spiked with exogenous compounds | 1 day
  measured (in %) by establishing difference plots between biochemical measurement results obtained for the CRMs and a panel of clinical specimens (see Clin Chem. 2018;64(3):455-464)
Non-commutability bias of certified reference materials (CRMs) consisting of frozen serum not spiked with exogenous compounds | 1 day
  measured (in %) by establishing difference plots between biochemical measurement results obtained for the CRMs and a panel of clinical specimens (see Clin Chem. 2018;64(3):455-464)
Non-commutability bias of external quality controls (EQA) consisting of Lyophilized serum spiked with exogenous compounds | 1 day
  Measured (in %) by establishing difference plots between biochemical measurement results obtained for the EQA and a panel of clinical specimens (see Clin Chem. 2018;64(3):455-464).
Non-commutability bias of external quality controls (EQA) consisting of Lyophilized serum not spiked with exogenous compounds | 1 day
  Measured (in %) by establishing difference plots between biochemical measurement results obtained for the EQA and a panel of clinical specimens (see Clin Chem. 2018;64(3):455-464).
Non-commutability bias of external quality controls (EQA) consisting of frozen serum spiked with exogenous compounds | 1 day
  Measured (in %) by establishing difference plots between biochemical measurement results obtained for the EQA and a panel of clinical specimens (see Clin Chem. 2018;64(3):455-464).
Non-commutability bias of external quality controls (EQA) consisting of frozen serum not spiked with exogenous compounds | 1 day
  Measured (in %) by establishing difference plots between biochemical measurement results obtained for the EQA and a panel of clinical specimens (see Clin Chem. 2018;64(3):455-464).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, PUPH, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - University Hospital Montpellier, Montpellier
  - University Hospital, Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided